CLINICAL TRIAL: NCT05293054
Title: Obsidian in Anastomotic Healing After Rectal Cancer Resection: A Prospective Clinical Feasibility Study
Brief Title: Healing of Rectal Anastomosis Sealed With a Concentrate Derived From the Patient's Blood, After Rectal Cancer Surgery
Acronym: OBANORES
Status: Completed | Type: Observational
Sponsor: University of Aarhus (Other)
Collaborators: Danish Cancer Society (Other)
Responsible Party: Sponsor
Other Study IDs: VEK: 1-10-72-187-20
Record Dates: First submitted 2022-02-28; First posted 2022-03-24 (Actual); Last update posted 2024-03-27 (Actual); Status verified 2024-03

CONDITIONS: Anastomotic Leak Rectum; Rectal Cancer; Anastomotic Leakage
MeSH Terms: conditions — Rectal Neoplasms; Anastomotic Leak | interventions — obsidian

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Application of autologous fibrin matrix (Obsidian) — When the patient is anaesthetized, 120 ml venous blood is collected for preparation of the autologous fibrin matrix. The blood is processed in the Vivostat® unit for 30 minutes making a 5-6 ml concentrate ready for application by use of a specific endoscopic kit device.
  When the rectal cancer resection is completed and the specimen is extracted, the Obsidian will be applied using minimal invasive technique and the endoscopic kit device.
  Step 1: 1.5-2ml. Obsidian is applied onto the rectal stump, with the circular stapler device inserted into the rectal stump. The circular stapler is then closed, but not yet fired.
  Step 2: 2.5-3ml Obsidian is applied 360 degrees around the anastomosis, while taking care not to increase tension on the anal intestine end. The circular stapler is then fired and removed. The water-air-leak test is performed according to standard clinical practice. Step 3: The remaining part of the Obsidian is then sealed 360 degrees around the anastomosis.

SUMMARY:
Rectal cancer is one of the most frequent cancer diseases, with more than 1500 new cases per year in Denmark. Fortunately, if the tumor is discovered early, surgeons can remove the part of the intestine that is afflicted, and they can often sew the intestine-ends back together, forming what is known as an anastomosis. However, in 10-15% of cases, this anastomosis doesn't heal completely, leading to anastomotic leakage. This is a serious complication, with detrimental effects for the individual patient. Previous measures to avoid this complication, have proven unsuccessful.

Obsidian is a mixture derived from the patients' own blood, that contains components of blood normally responsible for stopping bleeding and kickstarting the healing process. It is already used in other clinical settings and preliminary, yet unpublished, results from a pilot study have shown its promise in decreasing the risk of anastomotic leakage in rectal anastomosis. However, its use has not been examined when performing surgery for rectal cancer with minimally invasive technique, which is today's standard.

The main clinical hypothesis of this feasibility study is that it is possible for colorectal surgeons to apply Obsidian successfully on the anastomotic area with minimal invasive technique, as a supplement during rectal cancer resection with anastomosis.

This study will be conducted at the Department of Surgery, Aarhus University Hospital. 50 patients will be included, who will undergo minimally invasive rectal cancer surgery with an anastomosis. Right after the onset of anaesthesia, 120 ml of blood will be collected from the patient and will be processed, making a 5-6 ml Obsidian concentrate. When the tumor-bearing part of the rectum has been removed, Obsidian will be applied, according to a pre-specified protocol.

If the application is deemed successful (based on predefined assessment criteria) in at least 90% of our included patients, then this study will serve as a stepping stone for a bigger study, the aim of which will be to assess if this method can indeed bring down the rate of anastomotic leakage in such patients.

ELIGIBILITY:
Inclusion Criteria:

* Primary rectal cancer (adenocarcinoma) with the lower boarder within 15 cm from the anal verge assessed by rigid proctoscopy
* Clinical UICC stage I-III at time of rectal cancer diagnosis
* Deemed suitable for intended curative rectal cancer resection at MDT either by total mesorectal excision (TME) or partial mesorectal excision (PME)
* Scheduled for elective, minimal invasive surgery
* ECOG performance status 0-2
* Age at least 18 years
* Written and orally informed consent

Exclusion Criteria:

* Distant metastatic disease
* Locally advanced rectal cancer requiring extended resection
* Open surgery
* Benign lesions of the rectum
* Inflammatory bowel disease
* Another malignant disease within previous 2 years
* Inability and unwillingness to give informed consent
* Pregnant (positive pregnancy test) or breast feeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with biopsy proven rectal cancer subjected to minimally invasive rectal resection with anastomosis (TME or PME).
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2021-12-15 (Actual); Primary Completion 2023-11-08 (Actual); Study Completion 2023-11-08 (Actual)

PRIMARY OUTCOMES:
The rate of successful use and application of Obsidian as a supplemental procedure in the creation of rectal anastomosis with minimal invasive technique | This outcome is measured during the intervention.
  Defined as the surgeon being able re-inforce the anastomosis with Obsidian as described in our protocol. Assessment of the Obsidian application must be graded using the following rating assessment scale:
  'Complete'
  'Almost complete'
  'Incomplete'
  Each of these are detailed in the study protocol.
  To be able to view the use of Obsidian application as a successful method, then the application should be rated as 'Complete' or 'Almost complete' in at least 45 out of 50 (90%) patients.

SECONDARY OUTCOMES:
Time spent for creating a rectal anastomosis with application of Obsidian | This outcome is measured during the intervention.
  Time spent for creating the anastomosis with application of Obsidian is defined as: Time spent from inserting the circular stapler device in the rectal stump (Shortly before the start of Step 1 in Intervention Details), until the application around the circular anastomosis has been completed (End of Step 3 in Intervention Details).
The surgeon's self-assessment of the user-friendliness of using Obsidian | This outcome is measured immediately after the intervention.
  Surgeon's self-assessment of the user-friendliness of using Obsidian is graded in three grades: 1. Easy, 2. Difficult, but can be performed, 3. Very difficult
Anastomotic leak rate | Measured within 30 days after surgery
  Anastomotic leak is defined according to the definition as described by Rahbari NN.
Length of hospital stay | From, and including, day of surgery to, and including, day of discharge, or up to 90 days after surgery.
  Calculated as number of days
Re-hospitalization within 30 days after surgery | Measured within 30 days after surgery
  All re-hospitalizations at departments of any kind at hospitals in Central Denmark Region after surgery will be recorded, including reason for re-hospitalization.
Morbidity within 30 days after surgery graded ≥3 severity according to the Clavien-Dindo classification | Measured within 30 days after surgery
  Morbidity within 30 days after surgery include surgical and medical complications graded ≥2 severity according to the Clavien-Dindo classification, will be recorded.
  Surgical complications include bleeding, fascia dehiscence, ileus, surgical site infection, intra-abdominal abscess, and anastomotic leakage. Medical complications include cerebral complications (transitory ischemic attack, stroke), pulmonary complications (pneumonia, atelectasis, pleural effusion), cardiac complications (atrial fibrillation, acute myocardial infarction, heart failure), gastrointestinal complications (high stoma output, paralysis >4 days), urogenital complications (urinary tract infections, urinary retention, acute kidney insufficiency), thromboembolic complications (deep venous thrombosis, pulmonary embolism).
2-year mortality | Within 2 years after surgery
  For safety reasons, mortality within 2 years after surgery will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Lene H Iversen, DMSc, PhD, Principal Investigator — Department of Surgery, Aarhus University Hospital
Locations (1):
- Department of Surgery, Aarhus University Hospital, Aarhus, Central Jutland, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rahbari NN, Weitz J, Hohenberger W, Heald RJ, Moran B, Ulrich A, Holm T, Wong WD, Tiret E, Moriya Y, Laurberg S, den Dulk M, van de Velde C, Buchler MW. Definition and grading of anastomotic leakage following anterior resection of the rectum: a proposal by the International Study Group of Rectal Cancer. Surgery. 2010 Mar;147(3):339-51. doi: 10.1016/j.surg.2009.10.012. Epub 2009 Dec 11. PMID 20004450